CLINICAL TRIAL: NCT02657239
Title: Health Promotion and Disease Prevention Research Center
Brief Title: Mobility & Vitality Lifestyle Program
Acronym: MOVE UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven M. Albert, Principal Investigator, Chair of Department of Behavioral and Community Health Sciences, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1U48DP005001-01 (NIH)
Record Dates: First submitted 2015-11-25; First posted 2016-01-15 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Obesity
Keywords: Physical Function
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MOVE UP Intervention (Experimental): Subjects will participate in a healthy lifestyle weight management intervention focused on healthy eating and increasing physical activity
  Interventions: Behavioral: MOVE UP

INTERVENTIONS:
Behavioral: MOVE UP — Weight management behavioral program

SUMMARY:
MOVE UP is a weight management program for adults 60-75 in community settings led by trained community health workers.

DETAILED DESCRIPTION:
MOVE UP is a weight management program designed for adults who desire to lose weight and improve their overall health.

Topics include: Overall Health, Weight management, Healthy eating, Behavior change, Physical activity

ELIGIBILITY:
Inclusion Criteria:

1. Age 60-75 at time of program start
2. Self-reporting < 60 minutes per week of moderate structured physical activity
3. BMI >= 30 but < 40 for screen. In person measurement on site will allow for 27-45 as inclusion criteria.
4. Able to consent for participation and data collection
5. Medical release before start of Weight Management
6. Ability to walk with or without an assistive device
7. Can regularly attend sessions
8. Has not had bariatric surgery over the past year, or current use of weight loss prescription drug.

Exclusion Criteria:

1. Uncontrolled diabetes mellitus (FBS > 300 & A1C > 11%) [to be assessed by physician on medical release]
2. Uncontrolled hypertension (SBP > 180/110) %) [to be assessed by physician on medical release]
3. Recent hospitalization (past 6 months)
4. Active treatment for cancer (other than non-melanoma skin cancer)
5. Significant visual or hearing impairment
6. Dementia/psychiatric disorder
7. Inability to communicate in English/lack of translator

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery | 1 year
  Physical function objectively measured by Short Physical Performance Battery (SPPB) which includes gait speed, grip strength and chair stands, each ranked as 0-4 and summed for a total score of 0-12 units

SECONDARY OUTCOMES:
Self-reported Physical Function | 1 year
  Physical function self-reported with the MOS-SF36 - questions are assigned points for total points ranging fom 0-36
Weight | 1 year
  Weight in kilograms
Height | 1 year
  Height measured in meters
BMI | 1 year
  Calculated from objective measurements of height and weight above as weight in Kilograms divided height in meters-squared

CONTACTS AND LOCATIONS:
Overall Officials: Anne B. Newman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Community sites, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu X, King J, Boak B, Danielson ME, Boudreau RM, Newman AB, Venditti EM, Albert SM. Effectiveness of a behavioral lifestyle intervention on weight management and mobility improvement in older informal caregivers: a secondary data analysis. BMC Geriatr. 2022 Jul 28;22(1):626. doi: 10.1186/s12877-022-03315-w. PMID 35902809